CLINICAL TRIAL: NCT04587050
Title: Screening for Human Papillomavirus and Cervical Cancer in Young Women With Perinatally Acquired HIV
Brief Title: Screening for HPV and Cervical Cancer in Young Women With Perinatally Acquired HIV
Acronym: SHiP
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: 19SM5242
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: HIV Infections; Human Papillomavirus Infection; Cervical Cancer
Keywords: Cervical screening; HPV vaccination
MeSH Terms: conditions — HIV Infections; Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Serum blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Women with HIV sexually active: Women with perinatally acquired HIV aged 18 or over who are sexually active
  Interventions: Diagnostic Test: Human papillomavirus testing; Diagnostic Test: Cervical cytology; Diagnostic Test: HPV serology
- Cohort 2: Women with HIV not sexually active: Women with perinatally acquired HIV aged 18 or over who are not sexually active
  Interventions: Diagnostic Test: HPV serology

INTERVENTIONS:
Diagnostic Test: Human papillomavirus testing — HPV test from cervical sample using Cepheid GeneXpert HPV
  Groups: Cohort 1: Women with HIV sexually active
Diagnostic Test: Cervical cytology — Cervical cytology
  Groups: Cohort 1: Women with HIV sexually active
Diagnostic Test: HPV serology — HPV type specific serology (16/18) using ELISA from serum samples

SUMMARY:
This is a cross-sectional, observational study of high-risk HPV status, cervical cytology and HPV vaccine uptake and response in young women with perinatally acquired HIV.

DETAILED DESCRIPTION:
This is an observational study of cervical cytology assessment, high risk human papilloma virus (hr-HPV) status, and HPV antibody titres amongst adult women living with perinatally acquired HIV infection (PaHIV). Eligible consenting participants will have two samples taken; firstly, a cervical sample tested for cytology and Hr-HPV with the Cepheid GeneXpert HPV; secondly serum will be assessed for hr-HPV serology. All women with PaHIV, vaccinated and unvaccinated for HPV, over the age of 18 years will be eligible and will be recruited into one of two cohorts: (1) sexually active women: full study, cervical and blood sampling or (2) non-sexually active women, blood sampling only (total n=80). Follow up for abnormal smear results or hr-HPV positivity will be arranged through colposcopy.

ELIGIBILITY:
Inclusion Criteria - Cohort 1:

* Perinatally acquired HIV aged 18+
* Sexually active
* Able to give informed consent

Inclusion Criteria - Cohort 2:

* Perinatally acquired HIV aged 18+
* Able to give informed consent

Exclusion Criteria - Cohort 1:

* Pregnancy
* Not sexually active
* Previous total abdominal hysterectomy
* Unable to give informed consent

Exclusion Criteria - Cohort 2:

* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women living with perinatally acquired HIV aged 18 years or older
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tamara Elliott, Study Chair — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Opportunistic recruitment
Groups:
- Cohort 1: Women Living With HIV Who Are Sexually Active: Women with perinatally acquired HIV aged 18 or over who are sexually active
  Human papillomavirus testing: HPV test from cervical sample using Cepheid GeneXpert HPV
  Cervical cytology: Cervical cytology
  HPV serology: HPV type specific serology using ELISA from serum samples
- Cohort 2: Women Living With HIV Who Are Not Sexually Active: Women with perinatally acquired HIV aged 18 or over who are not sexually active
  HPV serology: HPV type specific serology using ELISA from serum samples
Period: Overall Study
Arm/Group | Cohort 1: Women Living With HIV Who Are Sexually Active | Cohort 2: Women Living With HIV Who Are Not Sexually Active
Started | 54 | 3
Completed | 54 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: Women Living With HIV Who Are Sexually Active: Women with perinatally acquired HIV aged 18 or over who are sexually active
  Human papillomavirus testing: HPV test from cervical sample using Cepheid GeneXpert HPV
  Cervical cytology: Cervical cytology
  HPV serology: HPV type specific serology (16/18) using ELISA from serum samples
- Cohort 2:Women Living With HIV Who Are Not Sexually Active: Women with perinatally acquired HIV aged 18 or over who are not sexually active
  HPV serology: HPV type specific serology (16/18) using ELISA from serum samples
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Women Living With HIV Who Are Sexually Active | Cohort 2:Women Living With HIV Who Are Not Sexually Active | Total
Number analyzed (Participants) | 54 | 3 | 57
Age, Customized [Count of Participants; unit: Participants]
  18-24 years | 22 | 2 | 24
  25+ years | 32 | 1 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 3 | 57
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White ethnicity | 5 | 1 | 6
  Black ethnicity | 20 | 1 | 21
  Other | 8 | 0 | 8
  Not stated | 21 | 1 | 22
Region of Enrollment [Number; unit: participants]
  United Kingdom | 54 | 3 | 57

OUTCOME MEASURES:

1. Primary Outcome: Prevalence of Abnormal Cervical Cytology
Description: Cervical sample taken in the clinic setting and sent to the laboratory for cytological examination. Prevalence of abnormal cytology is reported as the number of samples that had a non-normal cytology result (e.g. dyskaryotic cells) out of the total number tested
Time Frame: 1 year
Population: Zero women analysed in cohort 2 as these women were not sexually active and so cervical sample was not taken as per the protocol
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 2: Women Living With HIV Who Are Not Sexually Active: Women living with HIV who are not sexually active (no cervical sample taken)
Arm/Group | Cohort 1: Women Living With HIV Who Are Sexually Active | Cohort 2: Women Living With HIV Who Are Not Sexually Active
Number analyzed (Participants) | 46 | 0
Participants | 12 |

2. Secondary Outcome: Prevalence of High Risk HPV by Subtype
Description: Cervical sample taken in the clinic setting and tested for high-risk HPV on site using the Cepheid GeneXpert. Prevalence reported as the number of samples that were positive for any high-risk HPV out of all those tested
Time Frame: 1 year
Population: Zero samples analysed in cohort 2 as no cervical sample taken as these participants were not sexually active (as per protocol)
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1:Women Living With HIV Who Are Sexually Active: Women with perinatally acquired HIV aged 18 or over who are sexually active
  Human papillomavirus testing: HPV test from cervical sample using Cepheid GeneXpert HPV
  Cervical cytology: Cervical cytology
  HPV serology: HPV type specific serology using ELISA from serum samples
Arm/Group | Cohort 1:Women Living With HIV Who Are Sexually Active | Cohort 2: Women Living With HIV Who Are Not Sexually Active
Number analyzed (Participants) | 46 | 0
Participants
  HPV 16 | 2 |
  HPV 18/45 | 0 |
  Other high-risk HPV | 12 |
  Negative | 32 |

3. Secondary Outcome: Prevalence of CIN2+
Description: Participants with abnormal cytology and/or tested positive for high-risk HPV were referred for colposcopy. Prevalence reported as the number of participants who were diagnosed with CIN2+
Time Frame: 1 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1:Women With HIV Sexually Active: Women with perinatally acquired HIV aged 18 or over who are sexually active
  Human papillomavirus testing: HPV test from cervical sample using Cepheid GeneXpert HPV
  Cervical cytology: Cervical cytology
  HPV serology: HPV type specific serology using ELISA from serum samples
Arm/Group | Cohort 1:Women With HIV Sexually Active | Cohort 2: Women Living With HIV Who Are Not Sexually Active
Number analyzed (Participants) | 46 | 0
Participants | 1 |

4. Secondary Outcome: HPV Serology (16/18)
Description: Number of participants testing positive for HPV 16 and 18 antibodies out of the those tested
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Women Living With HIV Who Are Not Sexually Active: Women with perinatally acquired HIV aged 18 or over who are sexually active
  Human papillomavirus testing: HPV test from cervical sample using Cepheid GeneXpert HPV
  Cervical cytology: Cervical cytology
  HPV serology: HPV type specific serology using ELISA from serum samples
Arm/Group | Cohort 1: Women Living With HIV Who Are Not Sexually Active | Cohort 2: Women Living With HIV Who Are Not Sexually Active
Number analyzed (Participants) | 53 | 3
Participants
  HPV 16 positive serology | 44 | 1
  HPV 18 positive serology | 34 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No intervention
Groups:
- Cohort 2: Women With HIV Not Sexually Active: Women with perinatally acquired HIV aged 18 or over who are not sexually active
  HPV serology: HPV type specific serology using ELISA from serum samples
Arm/Group | Cohort 1:Women With HIV Sexually Active | Cohort 2: Women With HIV Not Sexually Active
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/3
Other Adverse Events (participants affected / at risk) | 0/54 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT04587050/Prot_SAP_000.pdf